CLINICAL TRIAL: NCT01021748
Title: A Phase I Study of Oral MK-2206 in Combination With Oral AZD6244 in Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: A Combination Therapy Study of MK-2206 and AZD6244 in Participants With Advanced Solid Tumors (MK-2206-010)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2206-010; 2009_698 (Other: Merck Registration Number)
Record Dates: First submitted 2009-11-25; First posted 2009-11-30 (Estimated); Results first posted 2018-08-07 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2017-11

CONDITIONS: Locally Advanced or Metastatic Solid Tumors
MeSH Terms: interventions — MK 2206; AZD 6244

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- MK-2206 45 mg QOD + AZD6244 75 mg QD (Experimental): Participants receive MK-2206 45 mg oral tablets once every other day (QOD) PLUS AZD6244 75 mg oral capsules once daily (QD) starting on Day 1 of each 28-day cycle.
  Interventions: Drug: MK-2206; Drug: AZD6244
- MK-2206 45 mg QOD + AZD6244 75 mg BID (Experimental): Participants receive MK-2206 45 mg oral tablets QOD PLUS AZD6244 75 mg oral capsules twice daily (BID) starting on Day 1 of each 28-day cycle.
  Interventions: Drug: MK-2206; Drug: AZD6244
- MK-2206 90 mg QW + AZD6244 50 mg BID (Experimental): Participants receive MK-2206 90 mg oral tablets once weekly (QW) PLUS AZD6244 50 mg oral capsules BID starting on Day 1 of each 28-day cycle.
  Interventions: Drug: MK-2206; Drug: AZD6244
- MK-2206 90 mg QW + AZD6244 75 mg QD (Experimental): Participants receive MK-2206 90 mg oral tablets QW PLUS AZD6244 75 mg oral capsules QD starting on Day 1 of each 28-day cycle.
  Interventions: Drug: MK-2206; Drug: AZD6244
- MK-2206 90 mg QW + AZD6244 75 mg BID (Experimental): Participants receive MK-2206 90 mg oral tablets QW PLUS AZD6244 75 mg oral capsules BID starting on Day 1 of each 28-day cycle.
  Interventions: Drug: MK-2206; Drug: AZD6244
- MK-2206 90 mg QW + AZD6244 100 mg QD (Experimental): Participants receive MK-2206 90 mg oral tablets QW PLUS AZD6244 100 mg oral capsules QD starting on Day 1 of each 28-day cycle.
  Interventions: Drug: MK-2206; Drug: AZD6244
- MK-2206 90 mg QW + AZD6244 150 mg QD (Experimental): Participants receive MK-2206 90 mg oral tablets QW PLUS AZD6244 150 mg oral capsules QD starting on Day 1 of each 28-day cycle.
  Interventions: Drug: MK-2206; Drug: AZD6244
- MK-2206 100 mg QW + AZD6244 100 mg QD (Experimental): Participants receive MK-2206 100 mg oral tablets QW PLUS AZD6244 100 mg oral capsules QD starting on Day 1 of each 28-day cycle.
  Interventions: Drug: MK-2206; Drug: AZD6244
- MK-2206 135 mg QW + AZD6244 100 mg QD (Experimental): Participants receive MK-2206 135 mg oral tablets QW PLUS AZD6244 100 mg oral capsules QD starting on Day 1 of each 28-day cycle.
  Interventions: Drug: MK-2206; Drug: AZD6244

INTERVENTIONS:
Drug: MK-2206 — Oral tablets
Drug: AZD6244 — Oral capsules
  Other Names: selumetinib

SUMMARY:
This study will investigate the safety and tolerability of combination therapy with MK-2206 and AZD6244 (selumetinib) and determine the maximum tolerated dose (MTD) and recommended Phase 2 dose (RPTD) for this drug combination in the treatment of participants with locally advanced or metastatic solid tumors. Preliminary efficacy data will also be collected.

The primary hypotheses for this study are that: 1) the Dose-limiting Toxicities (DLTs) observed in participants with locally advanced or metastatic solid tumors after administration of combination therapy with MK-2206 and AZD6244 will be dose-dependent and allow for identification of the MTD, and 2) oral administration of combination therapy with MK-2206 and AZD6244 to participants with advanced solid tumors will be generally well-tolerated.

ELIGIBILITY:
Inclusion Criteria:

* Participant has confirmed metastatic or locally advanced solid tumor that has failed to respond to standard therapy, progressed despite standard therapy, or therapies known to provide clinical benefit, or for whom efficacious standard therapy or any other therapy known to provide clinical benefit does not exist
* Participant has no history of prior cancer, except certain cervical, skin, or prostate cancers, or has undergone potentially curative therapy with no evidence of disease for 5 years
* At least 18 years of age
* Participant is able to swallow oral medications
* For participants enrolled in the MTD expansion cohorts, must have a diagnosis of Kirsten rat sarcoma viral oncogene homolog (KRAS) tumor-type non small-cell lung cancer (NSCLC). Additional tumor types (with specific mutations) may be added to the MTD expansion cohorts after discussion between Sponsor and Investigator

Exclusion Criteria:

* Participant has had chemotherapy, radiotherapy or biological therapy within 4 weeks of entering the study
* Participant is currently participating in or has participated in a study of an investigational compound or device within 30 days or 5x the compound's half-life of Cycle 1, Day 1
* Participant has known central nervous system metastases and/or carcinomatous meningitis
* Participant has a primary central nervous system tumor or spinal cord compression
* Participant is, at the time of signing informed consent, a regular user (including "recreational use") of any illicit drugs or had a recent history (within the last year) of drug or alcohol abuse
* Participant is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study
* Participant is human immunodeficiency virus (HIV) positive
* Participant is has history of hepatitis B or C or active hepatitis A
* Participant has a history or current evidence of heart disease
* Participant has uncontrolled high blood pressure
* Participant has poorly controlled diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2009-11-23 (Actual); Primary Completion 2012-11-26 (Actual); Study Completion 2014-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Tolcher AW, Khan K, Ong M, Banerji U, Papadimitrakopoulou V, Gandara DR, Patnaik A, Baird RD, Olmos D, Garrett CR, Skolnik JM, Rubin EH, Smith PD, Huang P, Learoyd M, Shannon KA, Morosky A, Tetteh E, Jou YM, Papadopoulos KP, Moreno V, Kaiser B, Yap TA, Yan L, de Bono JS. Antitumor activity in RAS-driven tumors by blocking AKT and MEK. Clin Cancer Res. 2015 Feb 15;21(4):739-48. doi: 10.1158/1078-0432.CCR-14-1901. Epub 2014 Dec 16. PMID 25516890

RESULTS

PARTICIPANT FLOW:
Groups:
- MK-2206 45 mg QOD + AZD6244 75 mg QD: Participants received MK-2206 45 mg oral tablets once every other day (QOD) PLUS AZD6244 75 mg oral capsules once daily (QD) starting on Day 1 of each 28-day cycle.
- MK-2206 45 mg QOD + AZD6244 75 mg BID: Participants received MK-2206 45 mg oral tablets QOD PLUS AZD6244 75 mg oral capsules twice daily (BID) starting on Day 1 of each 28-day cycle.
- MK-2206 90 mg QW + AZD6244 50 mg BID: Participants received MK-2206 90 mg oral tablets once weekly (QW) PLUS AZD6244 50 mg oral capsules BID starting on Day 1 of each 28-day cycle.
- MK-2206 90 mg QW + AZD6244 75 mg QD: Participants received MK-2206 90 mg oral tablets QW PLUS AZD6244 75 mg oral capsules QD starting on Day 1 of each 28-day cycle.
- MK-2206 90 mg QW + AZD6244 75 mg BID: Participants received MK-2206 90 mg oral tablets QW PLUS AZD6244 75 mg oral capsules BID starting on Day 1 of each 28-day cycle.
- MK-2206 90 mg QW + AZD6244 100 mg QD: Participants received MK-2206 90 mg oral tablets QW PLUS AZD6244 100 mg oral capsules QD starting on Day 1 of each 28-day cycle.
- MK-2206 90 mg QW + AZD6244 150 mg QD: Participants received MK-2206 90 mg oral tablets QW PLUS AZD6244 150 mg oral capsules QD starting on Day 1 of each 28-day cycle.
- MK-2206 100 mg QW + AZD6244 100 mg QD: Participants received MK-2206 100 mg oral tablets QW PLUS AZD6244 100 mg oral capsules QD starting on Day 1 of each 28-day cycle.
- MK-2206 135 mg QW + AZD6244 100 mg QD: Participants received MK-2206 135 mg oral tablets QW PLUS AZD6244 100 mg oral capsules QD starting on Day 1 of each 28-day cycle.
Period: Overall Study
Arm/Group | MK-2206 45 mg QOD + AZD6244 75 mg QD | MK-2206 45 mg QOD + AZD6244 75 mg BID | MK-2206 90 mg QW + AZD6244 50 mg BID | MK-2206 90 mg QW + AZD6244 75 mg QD | MK-2206 90 mg QW + AZD6244 75 mg BID | MK-2206 90 mg QW + AZD6244 100 mg QD | MK-2206 90 mg QW + AZD6244 150 mg QD | MK-2206 100 mg QW + AZD6244 100 mg QD | MK-2206 135 mg QW + AZD6244 100 mg QD
Started | 6 | 5 | 7 | 7 | 9 | 3 | 3 | 6 | 17
Treated | 6 | 4 (One participant was allocated, but not treated.) | 7 | 7 | 9 | 3 | 3 | 6 | 17
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not Completed | 6 | 5 | 7 | 7 | 9 | 3 | 3 | 6 | 16
Not completed — Adverse Event | 2 | 1 | 2 | 0 | 2 | 0 | 1 | 0 | 7
Not completed — Physician Decision | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 2
Not completed — Progressive Disease | 3 | 3 | 4 | 6 | 7 | 3 | 0 | 5 | 6
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Not Treated | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Baseline Analysis Population consisted of all participants who received at least one dose of study treatment.
Groups:
- MK-2206 45 mg QOD + AZD6244 75 mg QD: Participants received MK-2206 45 mg oral tablets QOD PLUS AZD6244 75 mg oral capsules QD starting on Day 1 of each 28-day cycle.
- MK-2206 45 mg QOD + AZD6244 75 mg BID: Participants received MK-2206 45 mg oral tablets QOD PLUS AZD6244 75 mg oral capsules BID starting on Day 1 of each 28-day cycle.
- MK-2206 90 mg QW + AZD6244 50 mg BID: Participants received MK-2206 90 mg oral tablets QW PLUS AZD6244 50 mg oral capsules BID starting on Day 1 of each 28-day cycle.
- Total: Total of all reporting groups
Arm/Group | MK-2206 45 mg QOD + AZD6244 75 mg QD | MK-2206 45 mg QOD + AZD6244 75 mg BID | MK-2206 90 mg QW + AZD6244 50 mg BID | MK-2206 90 mg QW + AZD6244 75 mg QD | MK-2206 90 mg QW + AZD6244 75 mg BID | MK-2206 90 mg QW + AZD6244 100 mg QD | MK-2206 90 mg QW + AZD6244 150 mg QD | MK-2206 100 mg QW + AZD6244 100 mg QD | MK-2206 135 mg QW + AZD6244 100 mg QD | Total
Number analyzed (Participants) | 6 | 4 | 7 | 7 | 9 | 3 | 3 | 6 | 17 | 62
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.0 (8.0) | 50.0 (5.9) | 48.9 (8.6) | 56.6 (7.3) | 56.1 (12.5) | 44.3 (8.0) | 63.0 (6.2) | 54.3 (15.3) | 64.7 (9.4) | 56.8 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 4 | 2 | 5 | 2 | 2 | 2 | 12 | 36
  Male | 2 | 1 | 3 | 5 | 4 | 1 | 1 | 4 | 5 | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Dose-limiting Toxicity (DLT)
Description: Adverse events (AEs) were graded using Common Terminology Criteria for Adverse Events (CTCAE), version 3.0. DLTs included: Grade 4 neutropenia lasting for ≥7 days; Grade 3 or Grade 4 neutropenia with fever >38.5ºC and/or infection requiring antibiotic or anti-fungal treatment; Grade 4 thrombocytopenia (≤25.0 x 10^9/L); Grade ≥3 non-hematologic toxicity with exceptions; Any drug-related AE, regardless of CTCAE Grade, leading to a dose modification of MK-2206 or AZD6244; Unresolved CTCAE Grade ≥3 drug-related toxicity requiring drug interruption for >14 days; ≥ Grade 3 signs or symptoms of glucose intolerance and accompanied by ≥ Grade 2 hyperglycemia (glucose >160 dL or 8.9 mmol/L); ≥ Grade 3 electrolyte abnormalities due to glucose intolerance and not attributable to another cause; Diagnosis of lactoacidosis or ketoacidosis; Persistent increases in corrected QT (QTc) interval (>60 msec from baseline and/or >500 msec); Clinically significant bradycardia.
Time Frame: Cycle 1 (Up to 28 days)
Population: The population consisted of all participants who completed ≥ 80% of the first cycle of combination therapy unless interruption of study medication was due to toxicity (e.g. DLT).
Measure: Number; unit: Participants
Arm/Group | MK-2206 45 mg QOD + AZD6244 75 mg QD | MK-2206 45 mg QOD + AZD6244 75 mg BID | MK-2206 90 mg QW + AZD6244 50 mg BID | MK-2206 90 mg QW + AZD6244 75 mg QD | MK-2206 90 mg QW + AZD6244 75 mg BID | MK-2206 90 mg QW + AZD6244 100 mg QD | MK-2206 90 mg QW + AZD6244 150 mg QD | MK-2206 100 mg QW + AZD6244 100 mg QD | MK-2206 135 mg QW + AZD6244 100 mg QD
Number analyzed (Participants) | 6 | 4 | 7 | 7 | 9 | 3 | 3 | 6 | 17
Participants | 0 | 2 | 2 | 1 | 3 | 0 | 2 | 0 | 3

2. Secondary Outcome: Number of Participants With a Tumor Response According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: Radiological evaluation (via computed tomography [CT] or magnetic resonance imaging [MRI]) of tumor response was assessed every 8 weeks post-treatment during Cycles 1-6, and per institutional standard of care in Cycle 7 and beyond. The best overall tumor response was the best response based on RECIST 1.1 recorded from the start of the study treatment until the end of treatment. Response categories included: Complete Response (CR): Disappearance of all target lesions; Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions; Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions; and Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. Participants whose tumor was not evaluable (NE) were missing a valid RECIST1.1 measurement at baseline. The best overall tumor response for participants is presented.
Time Frame: Baseline and after every 8 weeks of treatment until documentation of objective response or disease progression (Up to 2 years)
Population: The analysis population consisted of all participants with assessable disease at baseline or measureable disease at baseline per RECIST1.1.
Measure: Number; unit: Participants
Arm/Group | MK-2206 45 mg QOD + AZD6244 75 mg QD | MK-2206 45 mg QOD + AZD6244 75 mg BID | MK-2206 90 mg QW + AZD6244 50 mg BID | MK-2206 90 mg QW + AZD6244 75 mg QD | MK-2206 90 mg QW + AZD6244 75 mg BID | MK-2206 90 mg QW + AZD6244 100 mg QD | MK-2206 90 mg QW + AZD6244 150 mg QD | MK-2206 100 mg QW + AZD6244 100 mg QD | MK-2206 135 mg QW + AZD6244 100 mg QD
Number analyzed (Participants) | 6 | 3 | 7 | 7 | 9 | 3 | 2 | 6 | 13
Participants
  Complete Response | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Partial Response | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 2
  Stable Disease | 4 | 0 | 1 | 3 | 3 | 3 | 2 | 4 | 10
  Progressive Disease | 2 | 3 | 4 | 4 | 5 | 0 | 0 | 2 | 1

3. Primary Outcome: Number of Participants Who Experienced at Least One Adverse Event (AE)
Description: An AE was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of study drug, whether or not considered related to the use of the product. Any worsening of a pre-existing condition which was temporally associated with the use of study drug was also an AE. The number of participants who experienced at least one AE is presented.
Time Frame: Up to approximately 23 months
Population: The population consisted of all participants who received at least one dose of study treatment.
Measure: Number; unit: Participants
Arm/Group | MK-2206 45 mg QOD + AZD6244 75 mg QD | MK-2206 45 mg QOD + AZD6244 75 mg BID | MK-2206 90 mg QW + AZD6244 50 mg BID | MK-2206 90 mg QW + AZD6244 75 mg QD | MK-2206 90 mg QW + AZD6244 75 mg BID | MK-2206 90 mg QW + AZD6244 100 mg QD | MK-2206 90 mg QW + AZD6244 150 mg QD | MK-2206 100 mg QW + AZD6244 100 mg QD | MK-2206 135 mg QW + AZD6244 100 mg QD
Number analyzed (Participants) | 6 | 4 | 7 | 7 | 9 | 3 | 3 | 6 | 17
Participants | 6 | 4 | 7 | 7 | 9 | 3 | 3 | 6 | 17

4. Primary Outcome: Number of Participants Who Discontinued Study Treatment Due to an AE
Description: An AE was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of study drug, whether or not considered related to the use of the product. Any worsening of a pre-existing condition which was temporally associated with the use of study drug was also an AE. The number of participants who discontinued study treatment due to an AE is presented.
Time Frame: Up to approximately 20 months
Population: The population consisted of all participants who received at least one dose of study treatment.
Measure: Number; unit: Participants
Arm/Group | MK-2206 45 mg QOD + AZD6244 75 mg QD | MK-2206 45 mg QOD + AZD6244 75 mg BID | MK-2206 90 mg QW + AZD6244 50 mg BID | MK-2206 90 mg QW + AZD6244 75 mg QD | MK-2206 90 mg QW + AZD6244 75 mg BID | MK-2206 90 mg QW + AZD6244 100 mg QD | MK-2206 90 mg QW + AZD6244 150 mg QD | MK-2206 100 mg QW + AZD6244 100 mg QD | MK-2206 135 mg QW + AZD6244 100 mg QD
Number analyzed (Participants) | 6 | 4 | 7 | 7 | 9 | 3 | 3 | 6 | 17
Participants | 2 | 1 | 2 | 0 | 2 | 0 | 1 | 0 | 7

ADVERSE EVENTS:
Time Frame: Up to approximately 23 months
Description: The population consisted of all participants who received at least one dose of study treatment.
Arm/Group | MK-2206 45 mg QOD + AZD6244 75 mg QD | MK-2206 45 mg QOD + AZD6244 75 mg BID | MK-2206 90 mg QW + AZD6244 50 mg BID | MK-2206 90 mg QW + AZD6244 75 mg QD | MK-2206 90 mg QW + AZD6244 75 mg BID | MK-2206 90 mg QW + AZD6244 100 mg QD | MK-2206 90 mg QW + AZD6244 150 mg QD | MK-2206 100 mg QW + AZD6244 100 mg QD | MK-2206 135 mg QW + AZD6244 100 mg QD
Serious Adverse Events (participants affected / at risk) | 4/6 | 1/4 | 6/7 | 2/7 | 6/9 | 0/3 | 2/3 | 3/6 | 5/17
Other Adverse Events (participants affected / at risk) | 6/6 | 4/4 | 7/7 | 7/7 | 9/9 | 3/3 | 2/3 | 6/6 | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-2206 45 mg QOD + AZD6244 75 mg QD (N=6) | MK-2206 45 mg QOD + AZD6244 75 mg BID (N=4) | MK-2206 90 mg QW + AZD6244 50 mg BID (N=7) | MK-2206 90 mg QW + AZD6244 75 mg QD (N=7) | MK-2206 90 mg QW + AZD6244 75 mg BID (N=9) | MK-2206 90 mg QW + AZD6244 100 mg QD (N=3) | MK-2206 90 mg QW + AZD6244 150 mg QD (N=3) | MK-2206 100 mg QW + AZD6244 100 mg QD (N=6) | MK-2206 135 mg QW + AZD6244 100 mg QD (N=17)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Detachment of retinal pigment epithelium (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis C (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meningitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural fistula (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Complex partial seizures (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-2206 45 mg QOD + AZD6244 75 mg QD (N=6) | MK-2206 45 mg QOD + AZD6244 75 mg BID (N=4) | MK-2206 90 mg QW + AZD6244 50 mg BID (N=7) | MK-2206 90 mg QW + AZD6244 75 mg QD (N=7) | MK-2206 90 mg QW + AZD6244 75 mg BID (N=9) | MK-2206 90 mg QW + AZD6244 100 mg QD (N=3) | MK-2206 90 mg QW + AZD6244 150 mg QD (N=3) | MK-2206 100 mg QW + AZD6244 100 mg QD (N=6) | MK-2206 135 mg QW + AZD6244 100 mg QD (N=17)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (7)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arrhythmia supraventricular (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Auricular swelling (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amblyopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cataract subcapsular (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Detachment of macular retinal pigment epithelium (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Eye pain (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye swelling (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eyelid oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Macular fibrosis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Macular pigmentation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Maculopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ocular hypertension (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Periorbital oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal pigment epitheliopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scleral hyperaemia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (3) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 3 (8) | 3 (3) | 3 (7) | 3 (6) | 5 (6) | 3 (5) | 0 (0) | 2 (4) | 14 (20)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (6)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Faecal incontinence (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 5 (6) | 4 (5) | 1 (1) | 1 (1) | 2 (3) | 3 (3) | 8 (13)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophageal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 1 (2) | 1 (1) | 0 (0) | 5 (7) | 1 (1) | 0 (0) | 1 (2) | 3 (4)
Varices oesophageal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1) | 7 (10) | 4 (4) | 0 (0) | 0 (0) | 2 (4) | 3 (3) | 4 (4)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Axillary pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Fatigue (General disorders) | 3 (6) | 1 (1) | 4 (11) | 3 (4) | 3 (6) | 2 (4) | 1 (1) | 3 (4) | 11 (15)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 3 (7) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 7 (10)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Eyelid infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 4 (5)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nail injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (2) | 1 (7) | 1 (1) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (7)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 1 (3) | 0 (0) | 1 (3) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 4 (6)
Blood albumin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 1 (10) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood glucose increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Culture urine positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram T wave amplitude decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 4 (8)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brachial plexopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (2) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 5 (6)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Affective disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary hesitation (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal dryness (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergic cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 1 (2) | 2 (2) | 2 (4) | 3 (3)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 2 (3) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 4 (5)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 5 (10) | 4 (6) | 3 (5) | 1 (1) | 1 (1) | 2 (2) | 6 (10)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 2 (3) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 6 (8)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema annulare (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5)
Madarosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (4) | 1 (1) | 2 (2) | 1 (2) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 7 (9)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 6 (9) | 3 (8) | 3 (5) | 1 (1) | 5 (9) | 3 (7) | 1 (1) | 4 (13) | 9 (20)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (7)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (7)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Scab (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin erosion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission.